CLINICAL TRIAL: NCT01998581
Title: A Multicenter, Double-blind, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLBELLA® XC Injectable Gel for Lip and Perioral Enhancement
Brief Title: A Safety and Effectiveness Study of JUVÉDERM VOLBELLA® XC Injectable Gel for Lip and Perioral Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOLBELLA-004
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Subjects Desiring Lip Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JUVEDERM VOLBELLA® XC (Experimental): Lips injected with JUVEDERM VOLBELLA® XC
  Interventions: Device: JUVEDERM VOLBELLA® XC
- Restylane-L® (Active Comparator): Lips injected with Restylane-L®
  Interventions: Device: Restylane-L®

INTERVENTIONS:
Device: JUVEDERM VOLBELLA® XC — Up to 1.5 mL per lip (upper and lower) at each treatment (initial, touch-up, and repeat treatment). Additional product may be injected into the perioral area, as long as the total injection volume does not exceed 6.0 mL. Up to 6.0 mL allowed for repeat treatment.
  Arms: JUVEDERM VOLBELLA® XC
Device: Restylane-L® — Up to 1.5 mL per lip (upper and lower) at each treatment (initial, touch-up, and repeat treatment). Additional product may be injected into the perioral area, as long as the total injection volume does not exceed 6.0 mL.. Up to 6.0 mL allowed for repeat treatment.
  Arms: Restylane-L®

SUMMARY:
This is a multicenter, double-blind, randomized, controlled study of the safety and effectiveness of JUVÉDERM VOLBELLA® XC Injectable Gel versus Restylane-L® for lip and perioral enhancement.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Has a score of minimal, mild, or moderate on the LFS2, as agreed upon by the Treating and Evaluating Investigators, and desires at least 1 point of correction for one or both lips
* For treatment of perioral lines, has a POLSS score of severe or moderate as agreed upon by the Treating and Evaluating Investigators (all subjects are eligible for treatment in the vermilion body, oral commissures, vermilion border, Cupid's bow, and philtral columns)

Exclusion Criteria:

* Has lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
* Has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator
* Has undergone oral surgery (e.g., tooth extraction, orthodontia, or implantation) within 6 weeks before enrollment or is planning to undergo any of these procedures during the study
* Has ever undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
* Has undergone semipermanent dermal filler treatment (e.g., calcium hydroxylapatite, poly-L-lactic acid) in the lower face (below the orbital rim) within 24 months before enrollment or is planning to undergo such treatment during the study
* Has undergone temporary dermal filler treatment (e.g., hyaluronic acid or collagen) in the lower face (below the orbital rim) within 12 months before enrollment or is planning to undergo such treatment during the study
* Has undergone mesotherapy or cosmetic resurfacing (laser, photo-modulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) anywhere in the face or neck, or Botulinum toxin injections in the lower face (below the orbital rim) within 6 months before enrollment or is planning to undergo any of these procedures during the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- New Orleans, Louisiana, United States

REFERENCES:
- [Background] Geronemus RG, Bank DE, Hardas B, Shamban A, Weichman BM, Murphy DK. Safety and Effectiveness of VYC-15L, a Hyaluronic Acid Filler for Lip and Perioral Enhancement: One-Year Results From a Randomized, Controlled Study. Dermatol Surg. 2017 Mar;43(3):396-404. doi: 10.1097/DSS.0000000000001035. PMID 28157728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JUVEDERM VOLBELLA® XC | Restylane-L®
Started | 169 | 56
Completed | 123 | 44
Not Completed | 46 | 12
Not completed — Refused repeat treatment | 20 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Lost to Follow-up | 12 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Other reasons | 3 | 2
Not completed — Randomized but withdrew before treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Subject who received at least 1 treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | JUVEDERM VOLBELLA® XC | Restylane-L® | Total
Number analyzed (Participants) | 168 | 56 | 224
Age, Customized [Count of Participants; unit: Participants]
  <30 year | 7 | 1 | 8
  30 to 50 years | 57 | 17 | 74
  51 to 65 years | 88 | 33 | 121
  >65 years | 16 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 53 | 217
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Evaluating Investigator's Assessment of Lip Fullness on a 5-Point Scale
Description: Lip fullness is assessed by the Evaluating Investigator on the 5-point Lip Fullness Scale 2. Assessments range from 0=minimal flat or nearly flat contour, minimal red lip show (worse) to 4=very marked very significant red lip show, lower lip pout, and upper lip pout (best). A positive number change from baseline indicates improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Month 3
Population: Modified Intent-to-Treat: subjects who were randomized with a Lip Fullness Scale 2 baseline score of minimal, mild, or moderate and who received at least 1 treatment
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVEDERM VOLBELLA® XC | Restylane-L®
Number analyzed (Participants) | 165 | 53
Scores on a Scale
  Baseline | 1.2 (0.73) | 1.1 (0.70)
  Change from Baseline at Month 3 (N=152, 48): number analyzed (Participants) | 152 | 48
  Change from Baseline at Month 3 (N=152, 48) | 1.1 (0.75) | 1.0 (0.85)

2. Secondary Outcome: Percentage of Subjects in the JUVEDERM VOLBELLA® XC Treatment Arm With at Least a 1 Point Improvement From Baseline on the Perioral Lines Severity Scale (POLSS)
Description: The Evaluating Investigator evaluated the perioral lines severity using the 4-point POLSS where None=No lines; Mild=Few, shallow lines; Moderate=Some, moderate lines; and Severe=Many, deep lines or crevices. The percentage of subjects with at least a 1-point improvement is reported. In accordance with the analysis plan, the analysis with responder rate and 95% Confidence Interval was performed for the JUVEDERM VOLBELLA® XC group only.
Time Frame: Baseline, Month 3
Population: Subjects in the JUVEDERM VOLBELLA® XC group who received treatment in perioral lines with a baseline POLSS score of moderate or severe
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | JUVEDERM VOLBELLA® XC | Restylane-L®
Number analyzed (Participants) | 81 | 0
Percentage of Subjects | 65.9 [54.55 to 75.97] |

3. Secondary Outcome: Change From Baseline in Subject Satisfaction With Lips on the Lip Module of the FACE-Q Questionnaire
Description: Subjects evaluated satisfaction using the 22 items on the Satisfaction with Lip module of the FACE-Q questionnaire. Scores for each item are combined to create a scale ranging from 0 (worse) to 100 (best). A positive number in change from baseline indicates an improvement, and a negative number in change from baseline indicates a worsening.
Time Frame: Baseline, Month 3
Population: Modified Intent-to-Treat: subjects who were randomized with data at both time points and received at least 1 treatment
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | JUVEDERM VOLBELLA® XC | Restylane-L®
Number analyzed (Participants) | 153 | 51
Scores on a Scale | 37.6 [34.0 to 41.1] | 29.0 [21.9 to 36.0]

ADVERSE EVENTS:
Description: The Safety Population included subject who received at least 1 treatment. The Safety Population was used to assess adverse events and serious adverse events. Out of the safety population, 30 subjects were included in the JUVEDERM VOLBELLA® Repeat Treatment Arm for AE reporting.
  During the repeat treatment period, at the month 12 visit, JUVEDERM VOLBELLA® was administered regardless of the product used for initial treatment.
Groups:
- JUVEDERM VOLBELLA® XC Initial Treatment: Lips injected with JUVEDERM VOLBELLA® XC
- JUVEDERM VOLBELLA® Repeat Treatment: Lips re-injected with JUVEDERM VOLBELLA® XC
Arm/Group | JUVEDERM VOLBELLA® XC Initial Treatment | Restylane-L® | JUVEDERM VOLBELLA® Repeat Treatment
Serious Adverse Events (participants affected / at risk) | 5/168 | 1/56 | 0/30
Other Adverse Events (participants affected / at risk) | 85/168 | 28/56 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JUVEDERM VOLBELLA® XC Initial Treatment (N=168) | Restylane-L® (N=56) | JUVEDERM VOLBELLA® Repeat Treatment (N=30)
Non-Small Cell Lung Cancer Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Malignant Sweat Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JUVEDERM VOLBELLA® XC Initial Treatment (N=168) | Restylane-L® (N=56) | JUVEDERM VOLBELLA® Repeat Treatment (N=30)
Injection Site Mass (General disorders) | 54 | 15 | 12
Injection Site Bruising (General disorders) | 30 | 11 | 0
Injection Site Pain (General disorders) | 21 | 12 | 0
Injection Site Induration (General disorders) | 15 | 4 | 0
Injection Site Swelling (General disorders) | 14 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.